CLINICAL TRIAL: NCT00855478
Title: French Post-Marketing Surveillance Survey
Acronym: FR E-REGISTRY
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Early termination of patient enrollment based on business decision
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans Peter Stoll, MD, Cordis
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-FR-002
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2010-11-29 (Estimated); Status verified 2010-11

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Cypher drug-eluting stent
  Interventions: Device: Cypher stent ™ or Cypher Select ™

INTERVENTIONS:
Device: Cypher stent ™ or Cypher Select ™ — Cypher drug-eluting stent

SUMMARY:
To assess the safety and effecacy of the Cypher stent ™ & Cypher Select ™ in the normal use of medical practices, within the labeled indications.

DETAILED DESCRIPTION:
Multi-center, retrospective and prospective French register. This register does not impose any constraint on the evaluated population, the procedure, or the required examinations. The local practice routines should be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic ischemic heart disease due to de novo lesions (lesions <30 mm vessel reference diameter of 2.25 mm to 5 mm), assessed visually, native coronary arteries.

Exclusion Criteria:

* Patients suffering from coronary heart disease.
* Patients for whom treatment antiplatelet and / or anticoagulant is against the state;
* Patients with injuries incompatible with the full inflation of a balloon angioplasty;
* Transplant patients ;
* Patients with known allergy to Sirolimus, the stainless steel 316L, to polymethacrylates or copolymers polyolefins;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4080 (Actual)
Dates: Start 2006-05; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
There is no pre-specified endpoint. | 12 Months